CLINICAL TRIAL: NCT07191418
Title: Study-group on Palliative ERCP And RFA-ablation in Metastatic and Inoperable Pancreatic Tumors
Acronym: Spearmint
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Roberto Valente (Other Government)
Responsible Party: Sponsor-Investigator, Roberto Valente, MD, PhD, Senior Consultant Gastroenterologist, Region Västerbotten
Organization: Region Västerbotten (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Spearmint; CIV-23-03-042680 (Other: Swedish medical products agency)
Record Dates: First submitted 2025-09-08; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Pancreatic Cancer Metastatic to Liver
MeSH Terms: interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I: Endobiliary RFA + Biliary Stent Placement (Investigational Arm) (Experimental): Patients randomized to this arm will undergo:
  Endobiliary RFA Procedure:
  Performed via endoscopic retrograde cholangiopancreatography (ERCP). A radiofrequency ablation catheter, Habib™ EndoHPB is introduced into the biliary tract.
  Controlled thermal energy is applied to the malignant biliary stricture to ablate tumor tissue intraductally. RFA energy settings, duration of application, and number of applications will be standardized per protocol. Biliary Stent Placement: Immediately following RFA, a self-expandable metal stent (SEMS) or plastic stent will be deployed across the stricture to maintain biliary patency. The type and size of the stent will be based on clinical standard and anatomy.
  Supporting Treatment:
  Patients will receive standard systemic chemotherapy per national guidelines for metastatic pancreatic cancer (e.g., FOLFIRINOX or gemcitabine + nab-paclitaxel).
  Supportive care includes antibiotics peri-ERCP, analgesics, antiemetics, and biliary drainage monitoring.
  Interventions: Device: Habib™ EndoHPB; Procedure: ERCP
- Arm II: Biliary Stent Placement Alone (Control Arm) (Active Comparator): Patients randomized to the control group will receive:
  Biliary Stent Placement Only:
  Performed via ERCP as above, without RFA. A SEMS or plastic stent will be placed across the malignant stricture.
  Supporting Treatment:
  Identical systemic chemotherapy regimens and supportive care protocols as in Arm I.
  Interventions: Procedure: ERCP

INTERVENTIONS:
Device: Habib™ EndoHPB — This study will hold greater weight compared to previous ones, as it is randomized. It includes 178 patients, exclusively with pancreatic cancer, and is designed as a prospective investigation.
  Arms: Arm I: Endobiliary RFA + Biliary Stent Placement (Investigational Arm)
Procedure: ERCP — Endoscopic retrograde cholangiopancreatography (ERCP) as part of clinical routine.

SUMMARY:
Pancreatic ductal adenocarcinoma (PDAC) is a very aggressive cancer and may become the second leading cause of cancer death by 2030. About half of the patients are diagnosed late, when the cancer has already spread (mPDAC), and the outlook is very poor. Chemotherapy is currently the only treatment for mPDAC. It can slow the disease and slightly extend life, but usually only by a few months. There are no other treatments that clearly improve survival. Radiofrequency ablation (RFA) is a minimally invasive technique that uses high-frequency electrical energy to generate heat and destroy tumor cells. Radiofrequency energy raises the temperature of the tissue, leading to coagulative necrosis and tumor cell death. RFA is commonly used to treat certain types of cancer and pre-cancerous lesions, including liver, kidney, lung, and bone tumors. In addition to directly destroying tumor tissue, RFA may also enhance the immune system's ability to recognize and attack cancer cells by exposing tumor antigens that were previously hidden within the tumor mass. Most research on radiofrequency ablation (RFA) to date has focused on Barrett's esophagus and liver cancer. However, RFA is increasingly being explored in palliative care, where early results suggest potential benefits. Advances in miniaturized endoscopic technology have enabled the application of RFA in anatomically challenging locations, such as the bile duct. Studies, including case series and clinical trials, have demonstrated that RFA is both feasible and safe. However, its impact on overall survival remains uncertain. Many previous studies are limited by small sample sizes and heterogeneous populations, often including patients with different cancer types and disease stages, which introduces bias and limits the generalizability of findings. We have therefore designed a prospective study focusing on patients with bile duct obstruction due to pancreatic ductal adenocarcinoma (PDAC) with limited metastatic spread (oligometastatic mPDAC). This study aims to provide more robust evidence on the potential role of RFA in improving clinical outcomes in a carefully selected subset of patients with advanced PDAC.

DETAILED DESCRIPTION:
Pancreatic cancer is rapidly becoming a medical emergency. Its prognosis continues to worsen and it is projected to become the second leading cause of cancer-related deaths by 2030.

At diagnosis, approximately 50% of patients already present with metastatic disease (mPDAC). Despite advancements in chemotherapy and surgery, the overall prognosis for pancreatic cancer has remained largely unchanged over the past four decades. The incidence closely mirrors the mortality rate, indicating that most patients diagnosed with pancreatic cancer will ultimately succumb to local progression or distant metastasis. While nearly all patients with pancreatic cancer eventually enter a metastatic phase, there is a lack of innovative therapeutic options targeted to this population. In randomized controlled trials (RCTs), patients with mPDAC continue to have poor outcomes, even with current standard-of-care chemotherapy regimens such as FOLFIRINOX or gemcitabine plus nab- paclitaxel (GEM/nab-PTX), which yield a median overall survival (OS) of only 11.1 and 8.5 months, respectively. In contrast to PDAC, locoregional ablation therapies have increasingly become part of palliative care strategies for other cancers. Radiofrequency ablation (RFA) is a well- established technique that uses thermal energy to induce coagulative necrosis of tumor tissue.

It has demonstrated both curative and palliative benefits in various solid tumors. There is also emerging evidence that RFA may stimulate systemic anti-tumor immune responses, although these effects remain underexplored in pancreatic cancer. To date, only a few small studies have examined the role of localized ablation in PDAC, with limited insight into its survival benefits. However, recent advancements in endoscopic technology have made it possible to deliver RFA directly into the bile duct, even in anatomically challenging locations. The majority of PDAC tumors arise in the head of the pancreas, in close proximity to the bile duct. This frequently leads to compression or infiltration of the bile duct, and painless jaundice is often one of the first clinical signs. As the disease progresses, most patients develop biliary obstruction, requiring biliary decompression via endoscopic retrograde cholangiopancreatography (ERCP) or percutaneous transhepatic cholangiography (PTC).

During ERCP, RFA catheters small enough to pass through a duodenoscope can be used to deliver targeted ablation to tumor tissue involving the bile duct. Retrospective studies have suggested that intraductal RFA for malignant biliary obstruction may prolong survival in patients with a range of cancers, although these studies lack randomization and are often limited by heterogeneity and small sample sizes. To date, uncontrolled retrospective studies and a recent meta-analysis have suggested a potential survival benefit of radiofrequency ablation (RFA) in malignant biliary obstruction.

However, a recent randomized controlled trial (RCT) has questioned its true efficacy as an anti-cancer treatment.The majority of existing studies have focused on heterogeneous patient cohorts, often including mixed populations with malignant biliary strictures from both pancreatic and biliary tract cancers, and at various disease stages. As a result, it remains impossible to draw definitive conclusions regarding the survival benefit of RFA, due to subgroup underpowering and selection bias inherent in these study designs.

Moreover, robust data are lacking on several key endpoints, including cancer-specific survival, treatment safety, overall survival, and quality of life (QoL), all of which are essential for evaluating the clinical utility of RFA in this setting. In this trial, we aim to treat patients with metastatic pancreatic ductal adenocarcinoma (mPDAC) limited to liver-only metastases by delivering endoscopic radiofrequency ablation (RFA) directly into the bile duct. The primary objective is to apply ablative energy at the site where the primary pancreatic tumor infiltrates or compresses the bile duct, inducing partial tumor lysis via coagulative necrosis. Eligible patients must have a histologically or cytologically confirmed diagnosis of mPDAC and be undergoing palliative chemotherapy. Inclusion criteria target patients with a limited metastatic burden confined exclusively to the liver. Participants may have previously received biliary decompression through fully covered self-expandable metal stents (SEMS), plastic stents placed during ERCP, or internal/external percutaneous drainage (PTC). Additionally, patients with an established diagnosis of mPDAC on palliative chemotherapy who develop jaundice later in the disease course, such as those with tumors in the uncinate process, which may delay bile duct involvement due to anatomical considerations, will be included.

Patients will be randomized into two arms:

Control arm: placement of a fully covered metal stent alone Intervention arm: intraductal RFA followed by placement of a fully covered metal stent RFA within the bile duct is expected to ablate tumor tissue both inside and immediately outside the duct. Placement of the fully covered metal stent after RFA serves a prophylactic role, sealing any micro- or macroperforations caused by ablation and ensuring optimal bile flow management.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with newly diagnosed pancreatic cancer in the head of the pancreas causing compression on the bile duct.
* Metastatic stage to the liver
* Histologically or cytologically confirmed mPDAC.
* Cancer burden limited to maximum 5 metastases in the liver, each of them maximum 1 cm in the larger diameter.
* Patients must be under palliative chemotherapy treatment.
* Cancer should be radiologically measurable (in an area not previously irradiated).
* WHO performance status 0-2.
* Age 18-85 years.

Exclusion Criteria:

* Intellectual disability, unwillingness or language difficulties
* which hinders the ability to give informed consent.
* Ongoing extensive immunosuppression and/or severe leuko- or
* thrombocytopenia.
* Ongoing acute cholangitis.
* Ongoing sepsis.
* Acute kidney failure.
* Uncompensated heart failure or unstable coronary insufficiency
* (symptomatic/uncompensated).
* Pregnancy or breastfeeding.
* Any metastases outside the liver.
* Cardiac pacemakers/cardioverter defibrillators.
* Severe coagulopathy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint variable compares the Cancer Specific Survival between the two groups. | 6 months and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Umeå University Hospital, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: Undecided